CLINICAL TRIAL: NCT02535624
Title: Retroperitoneal Packing or Angioembolization for Hemorrhage Control of Pelvic Fractures - Quasi-randomized Clinical Trial of 56 Hemodynamically Unstable Patients With Injury Severity Score ≥ 33
Brief Title: Retroperitoneal Packing or Angioembolization for Hemorrhage Control of Pelvic Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Shandong Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PELVIC001
Record Dates: First submitted 2015-08-05; First posted 2015-08-28 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Shock, Hemorrhagic; Fractures, Bone; Multiple Trauma
MeSH Terms: conditions — Shock, Hemorrhagic; Fractures, Bone; Multiple Trauma | interventions — Drug Packaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ANGIO (Active Comparator): Patients with persistent hemodynamic instability (systolic blood pressure (SBP) <90 mmHg after the transfusion of 4 packed red blood cell (PRBC) units in the emergency department) were taken urgently to the angiography suite for pelvic angiography. These patients had to tolerate transfer to the suite. Patients receiving primarily angioembolization therapy were defined as the ANGIO group.
  Interventions: Procedure: ANGIO
- PACKING (Active Comparator): Indication for pelvic packing was persistent SBP<90 mmHg during the initial resuscitation period with 3000 ml of intravenous (IV) crystalloids and transfusion of 4 PRBC units. These patients were treated primarly with retroperitoneal packing, while angioembolization OR staff was unavailable (5pm-7am), and were defined as the PACK group.
  Interventions: Procedure: PACKING

INTERVENTIONS:
Procedure: PACKING — By retroperitoneal access the space in front of the pelvic fracture is compressed with surgical towels, which stops effectively venous bleeding
  Other Names: retroperitoneal pelvic packing
  Arms: PACKING
Procedure: ANGIO — Using en endovascular approach, bleeding arteries are identified and clotted using embolizing agents, or coils.
  Other Names: angioembolization
  Arms: ANGIO

SUMMARY:
This study is designed to answer whether minimal invasive vessel clotting (angioembolization) or open surgery (retroperitoneal packing) is more effective for pelvic fractures with massive bleeding. Patients admitted at daytime (7am-5pm) are treated with angioembolization while patients admitted at nighttime (5pm to 7am) are treated with open surgery.

DETAILED DESCRIPTION:
In patients with pelvic fracture uncontrollable bleeding is the major cause of death within the first 24h after injury. Early hemorrhage control is therefore vital for successful treatment. Nowadays, recommended techniques for hemorrhage control in pelvic fractures are retroperitoneal pelvic packing and angioembolization, dependent upon the available technical staff and resources and the condition of the patient.

Retroperitoneal pelvic packing, on the one hand, is a relatively simple method in controlling pelvic hemorrhage even with limited resources. Since 89% of pelvic fracture hemorrhage originates from venous bleeding, fracture stabilization and compressive hemostasis by packing is a reasonable approach. Angioembolization, on the other hand, has great high effectiveness with regard to bleeding control, but requires an angiography suite and technical staff. Since hemostasis of retroperitoneal venous bleeding often can be achieved by external pelvic fixation, angioembolization is required for the 11% arterial bleedings which are hard to control by packing. Even though many authors see both methods as complements, time is crucial in the multitrauma setting and the severely injured patient does not tolerate multiple interventions well. Until now good predictors for treatment choice are unavailable, and management of hemodynamically unstable pelvic fractures remains a matter of debate.

This study was designed to answer following questions:

* Is retroperitoneal pelvic packing or angiography superior with regard to in-hospital mortality, complications, required secondary procedures, or post-intervention blood loss?
* Which of these methods is the more rapid intervention in the acute setting?

ELIGIBILITY:
Inclusion Criteria:

* multitrauma defined as Injury Severity Score (ISS) > 17
* dislocated pelvic fracture type B or C according to Tile[10] on emergency department pelvic radiograph
* hemodynamic instability defined as systolic blood pressure (SBP) <90 mmHg after administration of 4 units of packed red blood cells (PRBC).

Exclusion Criteria:

* monotrauma, or ISS ≤ 17
* age > 65 years
* age < 18 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2003-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Number of participants deceased occurring in-hospital during or after treatment with packing or embolization | participants will be followed for the duration of hospital stay, an expected average of 6 weeks

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
Number of postoperative packed red blood cell units administered for each participant | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
Number of participants which required a secondary procedure (PACKING or ANGIO) after the primary intervention (PACKING or ANGIO) | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
  Packing for ANGIO and angioembolization for PACKING.
Time from admission (in minutes) to treatment (PACKING or ANGIO) for each participant | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
Procedural/surgical time (in minutes) for each participant | participants will be followed for the duration of hospital stay, an expected average of 6 weeks
Days on ICU for each participant | participants will be followed for the duration of hospital stay, an expected average of 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Zhou, MD, PhD, Study Director — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

REFERENCES:
- [Derived] Li Q, Dong J, Yang Y, Wang G, Wang Y, Liu P, Robinson Y, Zhou D. Retroperitoneal packing or angioembolization for haemorrhage control of pelvic fractures--Quasi-randomized clinical trial of 56 haemodynamically unstable patients with Injury Severity Score >/=33. Injury. 2016 Feb;47(2):395-401. doi: 10.1016/j.injury.2015.10.008. Epub 2015 Oct 22. PMID 26508436